CLINICAL TRIAL: NCT04022616
Title: Myeloid-Derived Suppressor Cell Function in Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, William Carson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-09142
Record Dates: First submitted 2019-06-15; First posted 2019-07-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Immediate Surgery: Adult patients with breast malignancy.
  Interventions: Other: Specimen collection
- Neo-adjuvant Chemotherapy: Adult patients with biopsy proven operable breast cancer who in the opinion of treating physician are suited to receive neo-adjuvant chemotherapy.
  Interventions: Other: Specimen collection
- Lymph Node Tissue: Adult patients with breast malignancy who will be having a primary lymph node removed during breast surgery.
  Interventions: Other: Specimen collection
- Metastatic Breast Cancer: Adult patients with biopsy proven stage IV breast cancer who are starting a new line palliative systemic therapy. A palliative systemic therapy will be defined in this trial as any chemotherapy regimen or combination of endocrine therapy with targeted agents such as cyclin dependent kinase 4/6 (CDK 4/6) inhibitors, HER2 targeting agents or inhibitors of mammalian target of rapamycin (mTOR).
  Interventions: Other: Specimen collection

INTERVENTIONS:
Other: Specimen collection — Specimens are obtained from patients who are being treated for breast malignancies.

SUMMARY:
Myeloid-Derived Suppressor Cell Function in Breast Cancer Patients

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to give informed consent
* Stage I-III breast malignancy

Exclusion Criteria:

* Unable to tolerate venipuncture

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being treated at the Ohio State Comprehensive Cancer Center and Stefanie Spielman Comprehensive Breast Center
Sampling Method: Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2010-06-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Isolate unfavorable immune cells MDSC from the peripheral blood or tumors of study subjects and test how strongly they inhibit function of favorable immune cells called Natural Killer Cells. | up to 1 year
  Function of Natural Killer Cells will be studied by measuring their ability to kill target cancer cells coated with monoclonal antibodies.
  isolate unfavorable immune cells called Myeloid Derived Suppressor Cells (MDSC) from the peripheral blood or the tumors of study subjects and test how strongly they inhibit function of favorable immune cells called Natural Killer Cells. Function of Natural Killer Cells will be studied by measuring their ability to kill target cancer cells coated with monoclonal antibodies.

SECONDARY OUTCOMES:
Isolate unfavorable immune cells called Myeloid Derived Suppressor Cells (MDSC) from the peripheral blood of study subjects who plan to start pre-operative chemotherapy for breast cancer to see if MDSC levels can predict who will respond to treatment. W | up to 1 year
  Percentage of MDSC at baseline and whether there is an association of baseline MDSC percent with response to chemotherapy.
Isolate unfavorable immune cells MDSC from peripheral blood of study subjects who receive pre-operative chemotherapy for breast cancer to identify changes in MDSC levels during treatment can predict who will respond to treatment. | up to 1 year
  Changes will be reported in percentage of MDSC and associations of such changes with response to chemotherapy.
Isolate lymph nodes from patients with breast cancer undergoing breast surgery to study what types of Natural Killer Cells are present. | up to 1 year
  Isolate a lymph nodes from patients with breast cancer undergoing breast surgery to study what types of Natural Killer Cells are present. Natural Killer cells are immune cells that are capable of killing cancer cells.

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, MD, Principal Investigator — Ohio State Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wesolowski R, Stiff A, Quiroga D, McQuinn C, Li Z, Nitta H, Savardekar H, Benner B, Ramaswamy B, Lustberg M, Layman RM, Macrae E, Kassem M, Williams N, Sardesai S, VanDeusen J, Stover D, Cherian M, Mace TA, Yu L, Duggan M, Carson WE 3rd. Exploratory analysis of immune checkpoint receptor expression by circulating T cells and tumor specimens in patients receiving neo-adjuvant chemotherapy for operable breast cancer. BMC Cancer. 2020 May 19;20(1):445. doi: 10.1186/s12885-020-06949-4. PMID 32429929
- See also: The Jamesline — http://cancer.osu.edu